CLINICAL TRIAL: NCT05904509
Title: The Relationship Between Insulin Resistance and Disease Severity and Duration in Atopic Dermatitis Patients
Brief Title: Insulin Resistance in Atopic Dermatitis Patients
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: E-54022451-050.05.04-56968
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; insulin resistance
MeSH Terms: conditions — Dermatitis, Atopic; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to determine the relationship between insulin resistance and disease duration and severity of atopic dermatitis.

DETAILED DESCRIPTION:
The aim of the study is to determine the relationship between insulin resistance and disease duration and severity of atopic dermatitis. EASI and SCORAD values and disease duration of atopic dermatitis patients are calculated during the examination. HOMA-IR blood test result is compared with the results.

ELIGIBILITY:
Inclusion Criteria:

* Atopic dermatitis patients confirmed by a dermatologist

Exclusion Criteria:

* patients younger than 2 years
* patients older than 80 years
* Atopic dermatitis patients without HOMA-IR result

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Atopic dermatitis patients confirmed by a dermatologist
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
HOMA-IR | 12 months
  Patients' blood test show the result of fasting insulin (microU/L) x fasting glucose (mmol/L)/22.5
SCORAD index | 12 months
  Severity scoring of atopic dermatitis is calculated for each patient in the study. 6 intensity items (erythema, edema/papulation, oozing/crusts, excoriations, lichenification, dryness); 2 subjective symptoms(itch, sleeplessness); body surface area are studied. Max score is 103.
EASI index | 12 months
  Eczema Area and Severity Index is calculated for each patient in the study. Body surface area, 4 intensity items(erythema, induration, excoriation, lichenification) are studied. Max score is 72.
Duration of the disease | 12 months
  The time from the first onset of symptoms of the disease to the present. The relationship between insulin resistance and disease duration is examined

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University Hospital, Istanbul, Turkey (Türkiye)